CLINICAL TRIAL: NCT06200909
Title: Caring for the Family Caregiver: Testing the Effect of Two Wellness Programs That Support the Well-being of Family Caregivers of Persons With Neurodegenerative Disorders
Brief Title: Self-Care Training for Family Caregivers of Persons With Neurodegeneration
Acronym: MCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Alexandra J. Fiocco, PhD, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2022-003
Record Dates: First submitted 2023-12-08; First posted 2024-01-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Caregiver Burden; Caregiver Stress
MeSH Terms: conditions — Caregiver Burden | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A prospective single-blinded mixed methods randomized controlled superiority trial, with participants randomized in blocks of 8-12 to either MM, PSY, or RC.
Who Masked: Outcomes Assessor
Masking Description: Researchers who engage in pre-post testing assessment will be blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Meditation (MM) (Experimental): 8-week mindfulness meditation program is based on Kabat-Zinn's MBSR program and will be led by MBSR-trained facilitators. The program has been modified to make it more accessible to caregivers. Weekly sessions will be 120-minutes long (instead of original 150-180-minute sessions). Formal meditation practices described in the original MBSR program (i.e., body scan, sitting meditation, mindful movement, mindful eating and walking) will be taught, in addition to loving kindness meditation (LKM). Participants will be given guided meditation recordings and compliance with home practice will be monitored with a practice log. The prescribed home practice has been modified to accommodate the needs of the caregiver: each practice is offered in 5- to 10-minute intervals (5 min, 10 min, and 20 min practice) to accommodate the caregiver's schedule.
  Interventions: Other: Mindfulness Meditation
- Psychoeducation (Active Comparator): Psychoeducation (PSY) condition will be similar to MM with respect to number and duration of weekly sessions and daily homework. PSY is a lecture-based program based on the "10 Keys"TM to Healthy Aging Course, an evidence-based program for older adults. Each session focuses on a specific topic related to wellness (e.g., nutrition, physical activity, medical screening) and caregiver-specific topics (e.g., understanding dementia and neurodegenerative disease, legal and financial issues).
  Interventions: Other: Psychoeducation
- Respite control (Active Comparator): Participant allocated to RC will not be exposed to a program, but will be offered 120-minutes of weekly respite care. Caregivers will be asked to record how they spend respite hours each week.
  Interventions: Other: Wait list control

INTERVENTIONS:
Other: Mindfulness Meditation — 8-week mindfulness meditation program, based on Kabat-Zinn's MBSR program and modified for caregivers. The intervention will be led by MBSR-trained facilitators.
  Arms: Mindfulness Meditation (MM)
Other: Psychoeducation — A lecture-style program based on the "10 Keys"TM to Healthy Aging Course, an evidence-based program for older adults. The program will be delivered by a facilitator experienced in delivering similar content.
  Arms: Psychoeducation
Other: Wait list control — Participants will receive two hours of respite from their caregiving responsibilities per week, for eight weeks. They will be given the opportunity to participate in either the MM or the PSY condition following completion of testing.
  Arms: Respite control

SUMMARY:
The purpose of this study is to assess whether an 8-week mindfulness program enhances psychological well-being (e.g., stress, depressive symptoms), biological indicators of stress (e.g., inflammation), and cognitive function (e.g., attentional ability) in primary family caregivers of persons with dementia or a related neurodegenerative disease. A total of 232 primary family caregivers aged 50+ years of age will be recruited for this study and randomized to one of three groups: mindfulness meditation (MM), psychoeducation (PSY) or caregiver respite (CR). All participants will complete three testing sessions: baseline (pre-intervention [T1]), post 8-week follow-up (post-intervention, [T2]), and 12-month follow-up (T3).

DETAILED DESCRIPTION:
The purpose of this study is to assess the benefits of 2 virtual self-care programs - mindfulness meditation or a psychoeducation support group - for family caregivers of persons with a neurodegenerative disorder. Both programs are 8-weeks in length. A third arm will include a respite-ony group, which may be considered "treatment as usual". Outcomes of interest include psychological well-being (e.g., stress, depressive symptoms), biological indicators of stress (e.g., inflammation), and cognitive function (e.g., attentional ability). All participants will complete three testing sessions: baseline (pre-intervention [T1]), post 8-week follow-up (post-intervention, [T2]), and 12-month follow-up (T3). The target sample is 232 family/informal caregivers, aged 50+ years old. All sessions will be conducted using the Zoom platform. Participants will be required to go to LifeLabs for blood collection. Blood results will be shared with participants.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age
* Currently a primary family caregiver
* Fluent in English

Exclusion Criteria:

* Existing mindfulness practice
* Diagnosed/Presenting with Post-traumatic Stress Disorder; Substance Disorder; Psychosis
* Unable to attend 8 sessions
* No access to a computer or high-speed internet
* Not willing to be randomized

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  10-item Likert-type scale that measured level of distress in the past month. The questionnaire will be modified to cover the past 2 weeks. Higher scores (range 0-40) indicate greater perceived stress.
Center for Epidemiological Studies - Depression | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  A 20-item Likert-type questionnaire that measures presence of depressive symptoms in the past week. Higher scores (range 0-60) indicate greater depressive symptoms.

SECONDARY OUTCOMES:
Zarit Burden Interview | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  A 22-item Likert-type scale that measures distress surrounding the caregiver role. Greater scores (range 0-88) indicate greater caregiver burden.
Flanker Task | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  The flanker task is a classic test of inhibitory control, in which participants are asked to indicate the direction in which a central arrow points while ignoring an array of "flanking" arrows. Flanker interference (difference in reaction times between congruent and incongruent trials for the correct responses, incongruent-congruent) will be calculated with greater scores indicating greater interference.
Allostatic Load Index | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up
  Blood samples will be collected to measure biomarkers of biological stress to create an allostatic load (AL) index. Using the count-based calculation method, biomarker values that fall above the 75th percentile of the sample distribution are categorized as 1 and those below the 75th percentile are categorized as 0; except for DHEA-S, HDL cholesterol, which are categorized as 1 for values that fall below the 25th percentile and 0 for values that fall above the 25th percentile (Seeman et al., 1997). Subsystem scores (metabolic, immune, cardiovascular, neuroendocrine) are created by summing the relative biomarker scores and a total AL index score is calculated by summing all biomarker scores. Greater AL index score indicates greater cumulative biological stress.

OTHER OUTCOMES:
Difficulties in Emotion Regulation - Short Form | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  A 16-item Likert-type scale that measure subjective, trait emotion-regulation ability. Participant respond to questions on a 5-point Likert scale with higher scores (range 16-80) indicating greater emotion dysregulation.
Five Factor Mindfulness Questionnaire - Short Form | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  A 24-item Likert-type questionnaire that measures the 5 facets of trait mindfulness. Subscale scores range from 8 to 40 for the observing, describing, acting with awareness, and non-judging facets, or 7 to 35 for the non-reacting facet, resulting in an overall FFMQ score range of 39 to 195. Higher scores indicate greater trait mindfulness.
Pearlin Mastery Scale | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  This 7-item scale measures the extent to which an individual regards their life chances as being under their personal control. Responses are given on a four-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree"
Self-Compassion Scale | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  26-item Likert type scale the measures self-compassion, with higher scores (range 1-5) indicating greater self-compassion.
WHO Quality of Life Scale - Brief | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  26-item questionnaire that measures satisfaction with quality of life, health and other areas of the respondent's life.Higher scores (range 0-100) indicate greater quality of life.
UMASS Stress Reduction Program Follow-up Questionnaire | Baseline, post-intervention (within 1 week following intervention completion), 12-month follow-up.
  Questionnaire to assess perceived change driven by participation in a stress reduction program. Will be administered to those in the psychoeducation and mindfulness condition only.
Fear and Resistance to Mindfulness Scale | Up to 1 week prior to participation in mindfulness condition; post-intervention (within 1 week following intervention completion)
  A 29-item scale designed to measure fears and resistances to engaging in mindfulness practice. Items are rated on a five-point Likert scale ranging from 1: Not at all like me to 5 (extremely like me). Will be completed by mindfulness condition only.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Fiocco, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified quantitative data will be posted on an open science framework when published in an open access journal. Data will also be made available upon request under ethical guidance.

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. J Psychopathol Behav Assess. 2016;38(3):443-455. doi:10.1007/s10862-015-9529-3
- [Background] Radloff LS. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1977;1(3):385-401. doi:10.1177/014662167700100306
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Juster RP, Bizik G, Picard M, Arsenault-Lapierre G, Sindi S, Trepanier L, Marin MF, Wan N, Sekerovic Z, Lord C, Fiocco AJ, Plusquellec P, McEwen BS, Lupien SJ. A transdisciplinary perspective of chronic stress in relation to psychopathology throughout life span development. Dev Psychopathol. 2011 Aug;23(3):725-76. doi: 10.1017/S0954579411000289. PMID 21756430
- [Background] Bohlmeijer E, ten Klooster PM, Fledderus M, Veehof M, Baer R. Psychometric properties of the five facet mindfulness questionnaire in depressed adults and development of a short form. Assessment. 2011 Sep;18(3):308-20. doi: 10.1177/1073191111408231. Epub 2011 May 17. PMID 21586480
- [Background] Pearlin LI, Lieberman MA, Menaghan EG, Mullan JT. The stress process. J Health Soc Behav. 1981 Dec;22(4):337-56. No abstract available. PMID 7320473
- [Background] Neff KD. The Development and Validation of a Scale to Measure Self-Compassion. Self and Identity. 2003;2(3):223-250. doi:10.1080/15298860309027
- [Background] Power MJ. Quality of life. In: Lopez SJ, Snyder CR, eds. Positive Psychological Assessment: A Handbook of Models and Measures. American Psychological Association; 2003:427-441. doi:10.1037/10612-027
- [Background] Gilbert P, Basran J, Plowright P, Matos M, Kirby J, Petrocchi N. Fears and Resistances to Mindfulness: Development of a Self-Report Scale. Mindfulness. 2023;14(11):2602-2616. doi:10.1007/s12671-023-02171-y